CLINICAL TRIAL: NCT03498573
Title: Evaluation of Minimally Invasive Alveolar Augmentation Procedure of Anterior Maxillary Ridge Using Tunneling Surgical Technique
Brief Title: Evaluation of Alveolar Augmentation Using Tunneling Surgical Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hussien Amer Elkady (Other)
Responsible Party: Sponsor-Investigator, Hussien Amer Elkady, dentist, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29004052103937
Record Dates: First submitted 2018-03-29; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Bone Atrophy
MeSH Terms: interventions — 1-methyl-1-piperidinomethane sulfonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tunneling surgical technique (Experimental)
  Interventions: Other: tunneling surgical technique

INTERVENTIONS:
Other: tunneling surgical technique — sticky bone prepared by centrifuge patient blood and mixing with xinograft
  Other Names: mpm

SUMMARY:
patients suffering from anterior maxillary horizontal bone defect the alveolar ridge will be augmented by minimally invasive tunneling technique utilizing MPM as bone graft and patients followed up for 14 weeks .

ELIGIBILITY:
Inclusion Criteria:

* Patients' age range from 18-60 years.
* Patients with horizontal bone defect in anterior maxillary area.
* Patients should be free from any systemic disease that may affect normal healing of bone and predictable outcome.

Exclusion Criteria:

• Patients with systemic diseases as history of radiation therapy or chemotherapy, hematological disorders and autoimmune diseases (may affect normal healing).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
bone formation | 14 weeks
  bone formation assessed by cone beam ct

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nevins ML, Camelo M, Nevins M, Schupbach P, Friedland B, Camelo JM, Kim DM. Minimally invasive alveolar ridge augmentation procedure (tunneling technique) using rhPDGF-BB in combination with three matrices: a case series. Int J Periodontics Restorative Dent. 2009 Aug;29(4):371-83. PMID 19639058